CLINICAL TRIAL: NCT02648269
Title: A Phase I Single Ascending Dose Safety, Pharmacokinetic and Pharmacodynamics Study of SEL-212 in Subjects With Elevated Blood Uric Acid
Brief Title: Safety and Pharmacodynamics of SEL-212 (Pegsiticase + SEL-110) in Subjects With Elevated Blood Uric Acid Levels
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Selecta Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEL-212/101
Record Dates: First submitted 2016-01-05; First posted 2016-01-07 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Gout
MeSH Terms: conditions — Gout

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SEL-110 (Experimental): Single intravenous dose of SEL-110
  Interventions: Drug: SEL-110; Biological: SEL-212
- SEL-212 (Experimental): Single intravenous dose of SEL-110 plus SEL-037 (pegsiticase)
  Interventions: Biological: SEL-212
- SEL-037 (Experimental): Single intravenous dose of SEL-037 (pegsiticase)
  Interventions: Biological: SEL-037

INTERVENTIONS:
Drug: SEL-110
  Arms: SEL-110
Biological: SEL-212
  Arms: SEL-110; SEL-212
Biological: SEL-037
  Arms: SEL-037

SUMMARY:
This Study will first evaluate the safety and pharmacokinetics of a single intravenous dose of SEL-110, a nanoparticle containing rapamycin, in subjects with elevated blood uric acid levels. This will be followed, in separate subjects, by evaluation of the safety, pharmacokinetics, pharmacodynamics and immunogenicity of a single intravenous dose of SEL-212, SEL-037 (pegsiticase) plus SEL-110, in subjects with elevated blood uric acid levels. Uricase is an enzyme that converts uric acid to the readily soluble allantoin that is then excreted and SEL-110 is designed to prevent unwanted anti-drug-antibodies (ADAs) from forming.

DETAILED DESCRIPTION:
This Study will first evaluate the safety and pharmacokinetics of a single intravenous dose of SEL-110, a nanoparticle containing rapamycin, in subjects with elevated blood uric acid levels. This will be followed, in separate subjects, by evaluation of the safety, pharmacokinetics, pharmacodynamics and immunogenicity of a single intravenous dose of SEL-212, SEL-037 (pegsiticase) plus SEL-110, in subjects with elevated blood uric acid levels. Uricase is an enzyme that converts uric acid to the readily soluble allantoin that is then excreted and SEL-110 is designed to prevent unwanted anti-drug-antibodies (ADAs) from forming. Cohorts of subjects in the SEL-110 only arms of the study will be given a single, ascending intravenous dose of SEL-110 and then monitored for safety and rapamycin levels (pharmacokinetics) over 30 days. Cohorts of subjects in the SEL-212 arms of the study will be given a single, ascending intravenous dose of SEL-110 with a fixed dose of SEL-037 and then monitored for safety, rapamycin levels, SEL-037 levels, uric acid levels and anti-drug-antibodies (ADAs) to SEL-037 for 30 days. One additional control group with receive a single intravenous infusion of SEL-037 at a fixed dose and then monitored for safety, SEL-037 levels, uric acid levels and anti-drug-antibodies (ADAs) to SEL-037 for 30 days

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ages 21 to 70 inclusive. Female subjects must be of non-childbearing potential;
* Has at the screening visit a serum uric acid ≥ 6 mg/dL, with or without a history of gout;
* The use of allopurinol, febuxostat (Uloric®), or probenecid as uric acid-lowering therapy is permissible if dosing has been stable for at least the month prior to the screening visit;
* Has adequate venous access and able to receive IV therapy;
* Evidence of a personally signed and dated informed consent document indicating that subject has been informed of all pertinent aspects of the study;

Exclusion Criteria:

* Prior exposure to any experimental or marketed uricase (for arms receiving SEL-037 or SEL-212);
* History of any allergy to pegylated products;
* Glucose-6-phosphate dehydrogenase deficiency or known catalase deficiency;
* History of hematological or autoimmune disorders, is immunosuppressed or immunocompromised;
* Presently taking a drug classified as CYP3A4 inducer or inhibitor;
* Has participated in a clinical trial within 30 days of the Screening;

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as assessed by frequency of drug related adverse events, graded by severity | 30 days
  To assess the safety and tolerability of a single infusion of SEL-110, SEL-212 or SEL-037 as assessed by frequency of drug related adverse events, graded by severity

SECONDARY OUTCOMES:
Pharmacokinetics of SEL-110 (AUC) | 30 days
  Measurement of the pharmacokinetics of SEL-110 over 30 days by area under the blood concentration versus time curve (AUC)
Pharmacokinetics of SEL-037 (AUC) | 30 days
  Measurement of the pharmacokinetics of SEL-037 over 30 days by area under the serum concentration versus time curve (AUC)
Pharmacodynamics of SEL-037 (blood uric acid levels) | 30 days
  Pharmacodynamics of SEL-037 by measurement of blood uric acid levels over 30 days
Immunogenicity of SEL-037 (measurement of anti-drug antibody levels) | 30 days
  Immunogenicity of SEL-037 by measurement of anti-drug antibody levels over 30 days

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - Miami Research Associates, Miami, Florida
  - Orlando Clinical Research Center, Inc., Orlando, Florida
  - SNBL Clinical Pharmacology Center Inc., Baltimore, Maryland
  - Davita Clinical Research, Minneapolis, Minnesota
  - Altoona Center for Clincal Research, Duncansville, Pennsylvania

REFERENCES:
- [Derived] Sands E, Kivitz A, DeHaan W, Leung SS, Johnston L, Kishimoto TK. Tolerogenic nanoparticles mitigate the formation of anti-drug antibodies against pegylated uricase in patients with hyperuricemia. Nat Commun. 2022 Jan 12;13(1):272. doi: 10.1038/s41467-021-27945-7. PMID 35022448